CLINICAL TRIAL: NCT04264390
Title: Piloting a Novel Home-based Telehealth Movement-to-music Program (M2M) for Increasing Physical Activity Among Adolescents With Cerebral Palsy: Protocol for a Randomized Controlled Trial
Brief Title: Piloting Home-based Movement-to-Music Among Adolescents With Cerebral Palsy: A Randomized Controlled Trial
Acronym: M2MCP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: American Academy of Cerebral Palsy and Developmental Medicine (Other)
Responsible Party: Principal Investigator, Byron Lai, Principle Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AACPDMJIA012001
Record Dates: First submitted 2020-02-07; First posted 2020-02-11 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Cerebral Palsy
Keywords: exercise; physical activity; telehealth
MeSH Terms: conditions — Cerebral Palsy; Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- M2M (Experimental): Participants will receive and be instructed to follow-along with 4 weeks of movement-to-music videos. Participants will also receive periodic behavioral coaching calls from a telecoach.
  Interventions: Behavioral: Movement-to-music
- Wait-list control (No Intervention): Participants will wait 4 weeks before starting the M2M program. Participants will be instructed to resume their normal daily activities during the wait-period.

INTERVENTIONS:
Behavioral: Movement-to-music — Movement-to-music is a physical activity program that was developed onsite at a state-of-the-art adapted fitness facility. The program includes movements that are coupled with music to enhance muscular strength, cardiorespiratory capacity, flexibility, and balance. For this study, the program will be packaged into playlists of exercise videos that will be given to participants. Participants will be instructed to complete the prescribed videos 3 times per week. Participants will also be asked to attend 4 behavioral coaching calls with a telecoach. The goals of the behavioral coaching calls will be to address issues with the technology components of the program and promote physical activity participation within the community and adherence to the movement-to-music videos.
  Other Names: M2M
  Arms: M2M

SUMMARY:
This study pilots the efficacy of a home-based movement-to-music program for increasing physical activity participation among adolescents with cerebral palsy. Half of the participants will receive the movement-to-music program immediately, which will include 4 weeks of exercise videos and periodic behavioral coaching calls. The other half of participants will wait 4 weeks before receiving the M2M program.

DETAILED DESCRIPTION:
The movement-to-music program has been tested among adults with physical disabilities and is currently being used in ongoing scale-up clinical trials. Current evidence suggests that the program can increase aspects of physical function among adults. The present study aims to test whether the same program can be used among adolescents with cerebral palsy. Study findings will be used to examine whether the videos require modifications prior to being implemented in a future scale-up trial for adolescents people with cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

1. Have a diagnosis of cerebral palsy
2. Be able to exercise with arms or be assisted through the movements by a parent
3. Be between the ages of 10-19 years
4. Have access to a Wi-Fi Internet connection at your home
5. Have access to a device that Is capable of viewing videos from YouTube (a television, computer tablet, laptop, or desktop)

Exclusion Criteria:

1. Does more than 60 minutes of moderate-to-vigorous physical activity per day in a normal week
2. Has complete blindness or deafness

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 59 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2021-09-07 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Changes in physical activity participation | Baseline and Week 4
  Participation in home, extracurricular, and community activities measured via the Children's Assessment of Participation and Enjoyment (CAPE). The CAPE is used to document changes in everyday activities outside of the school-setting. The CAPE provides 3 levels of scoring: 1) overall participation scores; 2) domain scores that reflect participation in formal and informal activities; and 3) scores that reflect participation in 5 types of activity (active, physical, recreation, social, skill-based, and self-improvement activities).

SECONDARY OUTCOMES:
Changes in Self-efficacy | Baseline and Week 4
  Exercise self-efficacy will be measured with the Exercise Self-Efficacy Scale (ESES). The ESES includes 8 items that assess an individual's perceived confidence in the ability to perform more than 40 min of moderate-intensity physical activity three times per week. The ESES is rated on a scale ranging from 0 (Not at all confident) to 100 (Completely confident). The scores are summed into a composite score that ranges between 0 and 100, where a higher score is indicative of a greater perceived level of confidence to participate in physical activity.
Changes in Goal-setting | Baseline and Week 4
  The EGS contains 10-items related to how an individual sets goals and plans exercise activities. Questions for each of the 2 subcategories (goal setting and planning) are scored on a 5-point scale ranging from 1 (does not describe) to 5 (describes completely). A higher score for the goal-setting subcategory reflects a greater skillset for setting and achieving goals. A higher score in the planning subcategory reflects a greater perceived ability to schedule exercise within the person's lifestyle.
Changes in Social support | Baseline and Week 4
  Social support will be measured by the Physical Activity Climate Questionnaire (PACQ), which was modified from a 12-item version of the questionnaire that demonstrated discriminant and convergent validity to assess physical activity climate among youth. The PACQ is a 15-item child-report measure of the perceived motivational 'climate' or autonomous support provided by the caregiver with regard to physical activity participation. Due to the nature of the questions, participants will be instructed to complete the PACQ without parental assistance. Questions are scored on a 7-point likert scale ranging from 1 (strongly disagree) to 7 (strongly agree). Higher average scores reflect a higher level of child-perceptions of autonomous support for physical activity behavior.
Changes in Outcome expectations | Baseline and Week 4
  Outcome expectations will be measured by the Multidimensional Outcomes Expectations for Exercise Scale (MOEES). The MOEES contains 15-items that assess three domains of outcome expectations, namely, physical, social, and self-evaluative outcome expectations. Questions are scored on a 5-point likert scale ranging from 1 (strongly disagree) to 5 (strongly agree) and totaled for each outcome expectation category.
Video Minutes Completed Throughout the Intervention (Adherence) | Week 1 through Week 4
  Adherence is defined as the number of movement-to-music video minutes completed throughout the program. The video minutes are objectively recorded via YouTube analytics. Participant's baseline characteristics will be regressed on video minutes, to explain who the program worked for.

OTHER OUTCOMES:
Changes in Perceived Pain | Baseline and Week 4
  Perceived pain will be measured via the National Institutes of Health Neuro-QoL Pediatric Pain short form.
Changes in Perceived Fatigue | Baseline and Week 4
  Perceived fatigue will be measured via the the National Institutes of Health Neuro-QoL Pediatric Fatigue short form.

CONTACTS AND LOCATIONS:
Overall Officials: Byron W Lai, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Children's Hospital of Alabama, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lai B, Vogtle L, Young R, Craig M, Kim Y, Gowey M, Swanson-Kimani E, Davis D, Rimmer JH. Telehealth Movement-to-Music to Increase Physical Activity Participation Among Adolescents With Cerebral Palsy: Pilot Randomized Controlled Trial. JMIR Form Res. 2022 Oct 28;6(10):e36049. doi: 10.2196/36049. PMID 36306154